CLINICAL TRIAL: NCT01931462
Title: A Single Arm Phase 1 Study of Microwave Coagulation Using 2450-MHz Antennae and CO2 Cooling in Partial Nephrectomy for T1 Renal Tumors
Brief Title: Microwave Coagulation in Partial Nephrectomy Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1080
Record Dates: First submitted 2013-08-23; First posted 2013-08-29 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Cancer of Kidney
Keywords: Cancer of the Kidney; Renal Cancer; Renal Neoplasms; Neoplasms, Kidney
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Certus 140™ (Experimental): During the operation: use of Certus 140™ microwave device for pre-coagulation of the kidney tissue adjacent to the tumor.
  Interventions: Device: Microwave pre-coagulation

INTERVENTIONS:
Device: Microwave pre-coagulation — The Certus 140™ system is used for microwave pre-coagulation of the tissue around the part of the kidney to be removed. This is done in place of the standard clamping to stop blood loss.

SUMMARY:
Partial nephrectomy (kidney removal) is a standard therapy for clinical T1 renal (kidney) tumors. The goals of surgery are to accurately remove the tumor with no cancer cells at the edge of the remaining tissue, to limit blood loss, and preserve kidney function. The most common technique is to clamp the blood supply to the entire kidney during removal and to surgically repair the tumor bed with suture and agents to stop bleeding. This stops the blood supply to the entire kidney including the healthy tissue, which can cause damage to the remaining tissue due to a shortage of oxygen if left clamped too long.

This study uses a microwave pre-coagulation technique using the Certus 140™ to facilitate a bloodless area near the tumor for accurate tumor removal and repair, while avoiding clamping the blood supply, but its effect on the function of kidney adjacent to tumor is unknown. If adequate stoppage of bleeding is achieved using the Certus 140™ with minimal heat spreading to the remaining tissue, clamping and a shortage of oxygen can be avoided.

The hypothesis is that microwave pre-coagulation is a safe method for providing the stoppage of bleeding during partial kidney removal.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a solitary, polar, clinical T1 renal mass
2. Patient must have adequate kidney function as measured by eGFR (estimated glomerular filtration rate) greater than or equal to 50 calculated from a standard care serum creatinine performed within 30 days prior to the partial nephrectomy operation.
3. Women of child-bearing potential must have negative serum or urine pregnancy test
4. Patient must be able to give written informed consent
5. Patient must be 18 years or older
6. No blood-thinning medications, including anti-inflammatory medications, herbs and supplements for at least 1 week prior to surgery

Exclusion Criteria:

1. T stage greater than clinical T1
2. Tumor extends beyond kidney into major veins, perinephric tissues, or adrenal gland
3. Prior surgery or radiation therapy to the region of interest
4. Patient has a single functioning kidney
5. Patient has an uncorrectable coagulopathy
6. Patient is not a surgical candidate due to underlying cardiac or other serious comorbid condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E Jason Abel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Certus 140™
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Certus 140™
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Effectiveness of Microwave Pre-coagulation Using the Certus 140™ System for Partial Nephrectomy on Renal Function Using the Estimated Glomerular Filtration Rate.
Description: We will be measuring the change in renal function as quantified by pre- and post-surgical estimated Glomerular Filtration Rate. Change = (6 week score - Baseline score)
Time Frame: 30 days prior to surgery (Baseline) and 6 weeks post surgery
Measure: Number; unit: estimated Glomerular Filtration Rate
Arm/Group | Certus 140™
Number analyzed (Participants) | 1
estimated Glomerular Filtration Rate
  Baseline | 66
  6 weeks post-surgery | 86
  Change from Baseline at 6 weeks | 20

2. Secondary Outcome: Blood Loss
Description: To assess the safety and efficacy of the Certus 140™ in establishing hemostasis by measuring blood loss. We will calculate the mean, median, standard deviation, and range of values for blood loss.
Time Frame: During the operation
Measure: Number; unit: mL
Arm/Group | Certus 140™
Number analyzed (Participants) | 1
mL | 300

3. Secondary Outcome: Operative Time
Description: To assess the safety and efficacy of the Certus 140™ in establishing hemostasis by measuring operative time. We will calculate the mean, median, standard deviation, and range of values for operative time.
Time Frame: During the operation
Measure: Number; unit: minutes
Arm/Group | Certus 140™
Number analyzed (Participants) | 1
minutes | 129

4. Secondary Outcome: Clamp Time
Description: To assess the safety and efficacy of the Certus 140™ in establishing hemostasis by measuring clamp time. We will calculate the mean, median, standard deviation, and range of values for clamp time.
Time Frame: During the operation
Population: This 1 subject was not clamped during the operation.
Measure: Number; unit: minutes
Arm/Group | Certus 140™
Number analyzed (Participants) | 1
minutes | 0

5. Secondary Outcome: Change in Renal Function
Description: To assess the safety and efficacy of the Certus 140™ in establishing hemostasis by measuring the change in renal function by nuclear scan and creatinine clearance. We will calculate the mean, median, standard deviation, and range of values for change in renal function by nuclear scan and creatinine clearance.
Time Frame: Within 30 days prior to operation and 6 weeks post operation
Measure: Number; unit: mg/dL (creatinine)
Arm/Group | Certus 140™
Number analyzed (Participants) | 1
mg/dL (creatinine)
  Baseline | 1.13
  6 weeks | 0.90

6. Secondary Outcome: Change in Functional Renal Volume
Description: To assess the safety and efficacy of the Certus 140™ in establishing hemostasis by measuring the change in functional renal volume as measured by MRI. We will calculate the mean, median, standard deviation, and range of values for change in functional renal volume as measured by MRI.
Time Frame: Within 30 days prior to operation and 6 weeks post-operation
Population: Subject renal volume not measured. Only normal/abnormal renal function was assessed.
Arm/Group | Certus 140™
Number analyzed (Participants) | 0

7. Secondary Outcome: Tumor Margin
Description: The percentage of subjects with tumor positive margins will be reported. Tissue pathology will occur during the operation and a final tissue pathology will be performed 6 weeks after the operation.
Time Frame: During the operation and 6 weeks post-operation
Measure: Number; unit: percentage with tumor positive margins
Arm/Group | Certus 140™
Number analyzed (Participants) | 1
percentage with tumor positive margins | 0

8. Secondary Outcome: Complication Rates
Description: Complication rates will be estimated using the methods of Kaplan and Meier.
Time Frame: During the operation
Measure: Number; unit: participants with complications
Arm/Group | Certus 140™
Number analyzed (Participants) | 1
participants with complications | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Certus 140™
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days